CLINICAL TRIAL: NCT01792505
Title: A Phase I Trial of Surgical Resection Followed by Vaccination With Dendritic Cells Pulsed With Tumor Lysate With Imiquimod for Patients With Malignant Glioma
Brief Title: Dendritic Cell Vaccine With Imiquimod for Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, John Yu, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19814
Record Dates: First submitted 2011-07-01; First posted 2013-02-15 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biological/Vaccine (Experimental)
  Interventions: Biological: Dendritic Cell Vaccine in combination with Imiquimod cream

INTERVENTIONS:
Biological: Dendritic Cell Vaccine in combination with Imiquimod cream — After a successful complete resection of malignant glioma, patients will receive a total of 3 vaccines, each are 2 weeks apart. Imiquimod cream will be applied prior to and after each vaccination.

SUMMARY:
Malignant gliomas are very aggressive and among the most common of brain tumors. A diagnosis carries with it a median survival of approximately 24 months. The current standard treatment of surgical resection followed by radiation therapy and chemotherapy has not substantially prolonged survival and even the few treatment options shown to exhibit small increases in survival primarily benefit certain (i.e., young) patient subpopulations.

Cancer vaccines represent one novel therapy for malignant gliomas. The goal is for the body to recognize the tumor cells are foreign and produce its own response to fight off recurring tumor cells. A promising means of causing an immune response so the body can create this immunity is through the use of dendritic cell (DC) vaccines.

DETAILED DESCRIPTION:
Dendritic cells are a small group of cells contained in everyone's white blood cell population. These cells are responsible for letting the immune system know that something foreign is in the body. Dendritic cells help the body ward off disease by alerting the immune system.

Imiquimod in an FDA-approved cream that is an immune response modifier, which will be used off-label in this study. Imiquimod cream (5%, 250 mg) will be self-applied topically by patients to a 4 x 5-cm outlined area of healthy skin overnight on days 1-5 of each cycle. Application and removal times will be recorded in treatment diaries. Dendritic cells will be injected intradermally into the imiquimod-treated site on day 3. Cycles will be repeated every 2 weeks for a total of three injections. This study will examine the effectiveness of using Imiquimod with DC vaccines, as previous studies within the oncology department have studied the effectiveness of DC vaccines.

Imiquimod (Aldara, 3M) is one of the better characterized imidazoquinolines and is the only one currently approved for clinical use as a topical ointment. It has been demonstrated to possess antiviral and antitumor properties, and it is approved for the treatment of genital warts. Vaccination studies in animal models have indicated that imidazoquinolines can boost the magnitude and quality of T cell responses. It is considered a Toll-like receptor agonist which controls the activation of dendritic cells.

In humans, it was shown that topical imiquimod treatment may enhance the immunogenicity of a melanoma vaccine. Additionally, injection of immature DCs into imiquimod-pretreated skin lead to DC activation in situ and enhanced migratory capacity to draining lymph nodes in cancer patients. In this study, the investigators test the safety and feasibility of imiquimod in a vaccine against brain cancer to induce a more potent immune response that what has previously been observed.

In prior Phase I and Phase II studies, patients who received chemotherapy following DC demonstrated longer progression free and overall survival than the patients who received DC or chemotherapy alone. The use of DC vaccines is considered investigational and has not yet been approved by the FDA, but the investigators have obtained an IND for use of the vaccines.

The purpose of this study is to determine whether after standard therapy of tumor resection surgery followed by DC vaccines with Imiquimod will not only generate (start) an immune response, but will provide longer progression-free survival. Subjects will have clinically indicated resection surgery and will consent to our screening study for vaccine trials (IRB #9225), under which subjects will have their tumor tissue analyzed in order to verify eligibility into this study.

Study procedures include the following: laboratory blood draws, urinalysis at screening, immunological testing, administration of the quality of life questionnaire, neurological exams, MRI testing, leukapheresis for dendritic cells, review of adverse events/concomitant medications.

Patients who were screened and not enrolled in this clinical trial due to screen failure will be notified of the reason for screen failure. Pre HIV counseling and appropriate referral resources will be provided. If the screen failure is due to the positive HIV test, appropriate post HIV counseling will be provided and appropriate referrals will be made. The charts of the patients with screen failures will be destroyed. The patients' charts who will be enrolled in the study will be kept in the locked cabinet in the research office. Patients will be assigned a unique identifying code known only to the research team. Data will be captured by various source documents, or, as necessary, abstracted from hospital medical records by an experienced registered nurse. The electronic data for viral testing will be accessible to research personnel only.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histopathological diagnosis of malignant glioma.
* Patients 18 years of age or older.
* Patients must have undergone maximal surgical resection of malignant glioma
* Both male and female of childbearing age entering the protocol must use a medically accepted form of birth control during the study, will be required to have a negative pregnancy test for female.
* Patients must have a Karnofsky performance score of at least 60%.
* Patients must be off steroids for at least two weeks prior to vaccination.
* Baseline hematologic and complete metabolic panel within one week of initiating therapy must fall within normal ranges
* Patient must be capable of signing IRB approved Research Consent and Release of Medical Records form.

Exclusion Criteria:

* Severe pulmonary, cardiac or other systemic disease associated with an unacceptable anesthetic or operative risk.
* The presence of an acute infection requiring active treatment will be criteria for delay or exclusion.
* Contraindication to MRI procedure unless otherwise determined by PI.
* Patients with a known history of an autoimmune disorder.
* Pregnancy.
* Patients positive for hepatitis B, hepatitis C, HIV I/II, syphilis, HTLV I/II, HCV.
* Patients with allergy to Gentamicin.
* Patient inability to participate as determined by PI discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-10; Primary Completion 2014-11-14 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
safety of an autologous tumor lysate- loaded dendritic cell (DC) vaccine with Imiquimod cream application | 1 year
  Safety relative to vaccine will be monitored in terms of Serious Adverse Events according to FDA regulations and recorded on a MedWatch 3500a form. A Data Safety Monitoring Committee will meet every 6 months to review AEs/SAE's. In the event of any subject death within a 30 day period following study agent administration, the DSMC will review the death within that time frame. If two deaths are deemed to be "probably" or "definitely' related to study agent administration, all study agent administrations will be stopped and the FDA and IRB will be notified of study cessation.

SECONDARY OUTCOMES:
progression free survival of patients after they receive tumor lysate-loaded DC vaccine with Imiquimod cream application. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Yu, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States